CLINICAL TRIAL: NCT03245268
Title: International BPA Registry
Status: Completed | Type: Observational
Sponsor: International CTEPH Association (Other)
Responsible Party: Sponsor
Other Study IDs: BPA Registry
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; CTEPH
Keywords: Balloon pulmonary angioplasty; BPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Balloon pulmonary angioplasty — BPA is an interventional technique where a balloon catheter is used to recanalize affected segments of pulmonary arteries identified during angiography.
  Other Names: BPA

SUMMARY:
The International Balloon Pulmonary Angioplasty (BPA) Registry is a prospective, multi-center, long-term observational project. Scheduled to start data collection in Q4 2017, the registry will run for approximately four years with a follow-up time for each patient of at least two years. Its primary objective is to investigate the efficacy and safety of BPA intervention in patients with chronic thromboembolic pulmonary hypertension (CTEPH) not amenable to pulmonary endarterectomy (PEA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with CTEPH according to the following criteria:

  * Mean PAP ≥ 25mmHg at rest; or if mean PAP < 25mmHg at rest, have exercise limitations from chronic thromboembolic disease
  * Abnormal ventilation perfusion lung scanning (VQ) scan, pulmonary angiogram, computer tomographic pulmonary angiogram, or magnetic resonance pulmonary angiogram confirming chronic thromboembolic disease as recommended by standard guidelines
* Treatment with anticoagulation for ≥ 3 months before diagnosis of CTEPH
* Naïve to BPA treatment
* Scheduled to undergo their first BPA session ≥ 1 day after enrollment. Enrollment is defined as date the consent is signed by the patient. Enrollment must occur before any BPA session
* Willing to provide informed consent

Exclusion Criteria:

* BPA treatment prior to enrollment
* Pulmonary hypertension cause other than World Health Organization (WHO) group IV (CTEPH)
* Targeted BPA treatment lesion other than from WHO group IV (CTEPH)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with CTEPH meeting the inclusion criteria listed below and scheduled to undergo BPA intervention are eligible for inclusion into the International BPA Registry.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by BPA-associated complications | Min. 2 years
Efficacy as assessed by change in PVR | Min. 2 years
  Change in pulmonary vascular resistance (PVR) from baseline to latest post-interventional follow-up hemodynamics
Efficacy as assessed by change in mPAP | Min. 2 years
  Change in mean pulmonary arterial pressure (mPAP) from baseline to latest post-interventional follow-up hemodynamics

SECONDARY OUTCOMES:
Compare volume of BPA cases across regions and case load at the end of recruitment | Min. 2 years
Analyze patient selection criteria for BPA across sites at the end of recruitment | Min. 2 years
At the end of follow-up, compare technical aspects of BPA as asssed by imaging modalities as used by the sites | Min. 2 years
  Imaging modalities encompass VQ scan, selective pulmonary angiogram, CT pulmonary angiogram, dual-energy CT, cone-beam CT, MRI, OCT and IVUS
At the end of follow-up, compare technical aspects of BPA as assessed by investigator-reported session goals | Min. 2 years
At the end of follow-up, compare technical aspects of BPA as assessed by number of sessions per patient and follow-up | Min. 2 years
At the end of follow-up, compare technical aspects of BPA as assessed by number of interventions per patient and follow-up | Min. 2 years
At the end of follow-up, compare technical aspects of BPA as assessed by technical limits | Min. 2 years
Analyze the use of PH targeted medical therapy before BPA | Min. 2 years
  PH targeted therapy will be categorised as prostacyclin, IP agonist, PDE5 inhibitor, ERA, guanylate cyclase stimulator and other
Analyze the use of PH targeted medical therapy after BPA | Min. 2 years
  PH targeted therapy will be categorised as prostacyclin, IP agonist, PDE5 inhibitor, ERA, guanylate cyclase stimulator and other
Analyze the impact of PH targeted medical treatment on key patient outcomes | Min. 2 years
  PH targeted therapy will be categorised as prostacyclin, IP agonist, PDE5 inhibitor, ERA, guanylate cyclase stimulator and other Key patient outcomes encompass WHO functional class, 6-minute-walk-distance, Borg dyspnoe score, haemodynamics and mortality
Health care resource use required to complete BPA | Min. 2 years
  As assessed by total hospital days in/out

CONTACTS AND LOCATIONS:
Overall Officials: Nick H Kim, Prof, Principal Investigator — International CTEPH Association
Locations (18):
- United States (5):
  - University of California San Diego, La Jolla, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
- University Clinics, Vienna, Austria
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- General University Hospital, Prague, Czechia
- France (2):
  - Centre Hospitalier Universitaire Grenoble-Alpes, Grenoble
  - L'Hôpital Marie Lannelongue, Le Plessis-Robinson
- Kerckhoff-Klinik GmbH, Bad Nauheim, Germany
- Japan (4):
  - National Hospital Organization Okayama Medical Center, Okayama
  - National Cerebral and Cardiovascular Center, Osaka
  - Keio University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
- VU Medical Center, Amsterdam, Netherlands
- European Health Center Otwock LLC, Warsaw, Poland
- Papworth Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Lang IM. Balloon Pulmonary Angioplasty for Chronic Thromboembolic Pulmonary Hypertension: Clinical Outcomes. Eur Cardiol. 2023 Apr 5;18:e11. doi: 10.15420/ecr.2022.29. eCollection 2023. PMID 37405334
- See also: Website of the International CTEPH Association — https://www.cteph-association.org/